CLINICAL TRIAL: NCT02091921
Title: Switch to Ticagrelor in Critical Limb Ischemia Anti-platelet Study
Acronym: STT-CLIPS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Leonardo Clavijo, Principal Investigator, Director, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: D5130L00068//ISSBRIL0198; HS-13-00562 (Other: IRB)
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Critical Limb Ischemia
Keywords: Critical Limb Ischemia, ticagrelor, Brilinta
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): All subjects will receive Ticagrelor.
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — All patients will be switched from clopidogrel to ticagrelor 90 mg twice daily for two weeks and the VerifyNow and VASP platelet reactivity assays repeated, samples will be collected before and 6±1 hours after the last ticagrelor dose.
  Other Names: Brilinta

SUMMARY:
Critical Limb Ischemia (CLI) is defined as limb pain that occurs at rest, or impending limb loss that is caused by severe compromise of blood flow to the affected extremity. CLI is a major cause of death and disability (secondary to myocardial infarction, stroke and amputation). The mortality in patients with CLI approaches 13-25% and 50% at one and five years respectively. High on-treatment platelet reactivity (HPR) in patients treated with aspirin and clopidogrel is associated with increased risk of recurrent cardiovascular events after percutaneous coronary interventions and coronary syndromes. Preliminary studies suggest that the prevalence of HPR in patients with critical limb ischemia treated with aspirin and clopidogrel is as high a 78.5%. In patients with coronary artery disease ticagrelor overcomes non-responsiveness to clopidogrel. However, the antiplatelet effect of ticagrelor in patients with critical limb ischemia is unknown.

DETAILED DESCRIPTION:
Study Aim: This pilot study aims to investigate platelet function after switching from clopidogrel to ticagrelor in patients with critical limb ischemia.

Fifty patients with diagnosis of CLI (Rutherford class IV-VI) treated with clopidogrel 75 mg and aspirin 81 mg daily will be tested for inhibition of platelet aggregation using the VerifyNow P2Y12 and VASP assays before and 6±1 hours after their daily clopidogrel dose. All patients will then be switched from clopidogrel to ticagrelor 90 mg twice daily for two weeks and the VerifyNow and Vasodilator-Stimulated Phosphoprotein (VASP) platelet reactivity assays repeated, samples will be collected before and 6±1 hours after the last ticagrelor dose. For exploratory analysis, patients will be divided in two groups based on the P2Y12 reaction units (PRU): Group 1. High on treatment platelet reactivity on clopidogrel (HPR), defined as P2Y12 reaction units (PRU) ≥208 and Group 2. Appropriate platelet inhibition on clopidogrel (API), defined as P2Y12 reaction units (PRU) <208. If subjects are withdrawn from the study prior to completion due to the high co-morbidity rate of this population, additional subjects will be enrolled to reach a total of 50 completed subjects for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of CLI (Rutherford class IV, V and VI) on continuous dual antiplatelet therapy with aspirin 81 mg and clopidogrel 75 mg daily for at least 14+2 days .

Exclusion Criteria:

* Chronic use of nonsteroidal anti-inflammatory drugs, thrombocytopenia (platelet count <100 × 103/μl), hemoglobin <10 g/dL, use of an oral anticoagulant (warfarin) or low molecular weight heparin within 14 days, GPIIb/IIIa inhibitors, or fibrinolytic drugs within 30 days. Pregnancy, <18 or >80 years of age, current smoking (>1 pack per day), concomitant therapy with strong cytochrome P450 3A inhibitors or inducers within 14 days, concomitant antithrombotic therapy other than aspirin within 14 days, hypercoaguable states. History of medication non-compliance, drug or alcohol abuse within 2 years. Acute coronary syndrome or coronary drug-eluting stenting within 1 year. Peripheral vascular revascularization procedures (surgical or endovascular) and/or amputation within one month. Contraindications for ticagrelor including: hypersensitivity to ticagrelor or any of the excipients, Active pathological bleeding, History of intracranial hemorrhage and Severe hepatic impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-02-16 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Clavijo, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with diagnosis of CLI (Rutherford class IV, V and VI) on continuous dual antiplatelet therapy with clopidogrel 75 mg and aspirin 81 mg daily for at least 14+2 days
Pre-assignment Details: A total of 53 patients consented and enrolled the study. 3 patients were excluded from the study and did not complete the study; one developed a skin reaction after the first IP dose; the other two due to events unrelated to the study (Pneumonia and Rheumatoid arthritis pericarditis).
  50 Patients completed the study.
Period: Overall Study
Arm/Group | Experimental
Started | 53
Completed | 50
Not Completed | 3
Not completed — Adverse Event | 3

BASELINE CHARACTERISTICS:
Population: The study analysis was based on the 50 patients who completed the study
Units Other Than Participants: blood samples
Arm/Group | Experimental
Number analyzed (Participants) | 50
Number analyzed (blood samples) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: To Determine Platelet Inhibition Before and After Switching for Two Weeks From Clopidogrel to Ticagrelor in Patients With CLI.
Description: Patients platelet inhibition was analyzed based on the P2Y12 reaction units (PRU) as high on treatment platelet reactivity (HPR), defined as P2Y12 reaction units (PRU) ≥208 and appropriate platelet inhibition on (API), defined as P2Y12 reaction units (PRU) <208
Time Frame: Two weeks
Measure: Mean (95% Confidence Interval); unit: P2Y12 reaction units (PRU)
Groups:
- Ticagrelor: All patients were switched from clopidogrel to ticagrelor 90 mg twice daily for two weeks
Arm/Group | Ticagrelor
Number analyzed (Participants) | 50
P2Y12 reaction units (PRU)
  Clopidogrel Baseline | 173 [149 to 196]
  Clopidogrel 6+-1 hour after the baseline dose | 140 [116 to 163]
  Ticagrelor Baseline | 71 [47 to 94]
  Ticagrelor 6+-1 hour after baseline | 63 [39 to 86]

2. Secondary Outcome: Establish the Number of Participants in the High On-treatment Platelet Reactivity (HPR) on Clopidogrel Group Who Demonstrated Appropriate Platelet Inhibition (API) After Switching to Ticagrelor for Two Weeks.
Description: This measure was obtained by the number of participants who demonstrated high on treatment platelet reactivity (PRU > / = 208) on Clopidogrel, and the number of participants who also resulted in the Appropriate Platelet Inhibition (PRU < 208) after switching to Ticagrelor for two weeks of uninterrupted therapy x 100% .
Time Frame: Two weeks
Population: Participants who demonstrated on the High Platelet Reactivity (HPR) on clopidogrel and had Appropriate Platelet Inhibition (API) on ticagrelor
Measure: Count of Participants; unit: Participants
Groups:
- HPR on Clopidogrel and API on Ticagrelor: Participants who demonstrated HPR on clopidogrel
Arm/Group | HPR on Clopidogrel and API on Ticagrelor
Number analyzed (Participants) | 18
Participants | 17

3. Secondary Outcome: Establish the Number of Participants With Appropriate Platelet Inhibition on Clopidogrel Who Demonstrated Appropriate Platelet Inhibition After Switching to Ticagrelor for Two Weeks.
Description: The measure was obtained from the number of participants in the Appropriate Platelet Inhibition (PRU < 208) on Clopidogrel and who remained with Appropriate Platelet Inhibition after switching to Ticagrelor for two weeks of uninterrupted therapy x 100
Time Frame: Two weeks
Population: Participants who demonstrated API on Clopidogrel and remained with API after switching to Ticagrelor
Measure: Count of Participants; unit: Participants
Groups:
- API on Clopidogrel and API on Ticagrelor: Participants with Appropriate Platelet Inhibition (API) on Clopidogrel.
Arm/Group | API on Clopidogrel and API on Ticagrelor
Number analyzed (Participants) | 32
Participants | 32

4. Secondary Outcome: Evaluate the Correlation Between PRU and VASP-PRI in CLI Patients During Clopidogrel Versus Ticagrelor Antiplatelet Therapy.
Description: Correlation between the P2Y12 Reaction Units (PRU) and the Vasodilator-Stimulated Phosphoprotein Assay-Platelet Reactivity Index (VASP-PRI) used to test the inhibition of platelet aggregation after two weeks of uninterrupted therapy with Clopidogrel versus Ticagrelor in CLI participants
Time Frame: Two weeks
Population: All participants were on Clopidogrel 75mg daily for at least two weeks and then switched to Ticagrelor 90mg twice daily for two weeks of uninterrupted therapy
Measure: Number; unit: Correlation Coefficient
Units Other Than Participants: Correlation Coefficient
Groups:
- Correlation of PRU and VASP-PRI: Participants who were switched from clopidogrel to ticagrelor
Arm/Group | Correlation of PRU and VASP-PRI
Number analyzed (Participants) | 50
Number analyzed (Correlation Coefficient) | 200
Correlation Coefficient
  Clopidogrel | 0.73
  Ticagrelor | 0.47
  Overall Group | 0.6

ADVERSE EVENTS:
Time Frame: Two weeks
Description: The adverse event and/or serious adverse event, used to collect adverse event information, adheres to the clinicaltrials.gov definition
Groups:
- Experimental: All participants will switch from clopidogrel to ticagrelor for two weeks
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 1/53
Other Adverse Events (participants affected / at risk) | 1/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=53)
Hospitalization for Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — considered unrelated to the study intervention
Rheumatoid arthritis pericarditis (Immune system disorders) | 1 (1) — considered unrelated to the study intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=53)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes